CLINICAL TRIAL: NCT07114601
Title: A Phase 1a/b Multicenter, Open-Label Trial to Evaluate Safety, Tolerability, and Dosimetry of LY4257496, a GRPR-Targeted Radioligand Therapy, in Adults With GRPR-Positive Advanced Solid Tumors (OMNIRAY)
Brief Title: A Study of LY4257496 in Participants With Cancer (OMNIRAY)
Acronym: OMNIRAY
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27354; J6C-OX-JKFA (Other: Eli Lilly and Company); 2025-522367-15-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-30; First posted 2025-08-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Breast Neoplasms; Colorectal Neoplasms; Prostate Neoplasm; Endometrial Neoplasms; Neoplasm Metastasis
Keywords: GRPR-positive
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Endometrial Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- LY4257496 Phase 1a Dose Escalation (Cohort A1) (Experimental): LY4257496 administered intravenously (IV)
  Interventions: Drug: LY4257496; Diagnostic Test: LY4257529
- LY4257496 Phase 1a Dose Optimization (Cohort A2) (Experimental): LY4257496 administered IV
  Interventions: Drug: LY4257496; Diagnostic Test: LY4257529
- LY4257496 + Standard of Care Phase 1b Cohort B (Experimental): Tumor specific cohort will receive LY4257496 alone or with standard of care anticancer therapy(ies)
  Interventions: Drug: LY4257496; Drug: Standard of Care Anticancer Therapies; Diagnostic Test: LY4257529
- LY4257496 Phase 1b Cohort C (Experimental): Tumor specific cohort will receive LY4257496
  Interventions: Drug: LY4257496; Diagnostic Test: LY4257529
- LY4257496 Phase 1b Cohort D (Experimental): Tumor specific cohort will receive LY4257496
  Interventions: Drug: LY4257496; Diagnostic Test: LY4257529

INTERVENTIONS:
Drug: LY4257496 — Administered IV
Drug: Standard of Care Anticancer Therapies — Fulvestrant, Imlunestrant, Aromatase Inhibitors, Capecitabine, Abemaciclib
  Arms: LY4257496 + Standard of Care Phase 1b Cohort B
Diagnostic Test: LY4257529 — Administered IV at select sites

SUMMARY:
The main purpose of this study is to evaluate safety, tolerability, and efficacy of LY4257496 alone and as part of relevant standard of care (SOC) combination therapy in participants with Gastrin-releasing Peptide Receptor (GRPR)-positive advanced breast, colorectal, prostate, and endometrial cancer. The study will also evaluate the safety, tolerability, and efficacy of LY4257529 to identify cancer with high levels of a protein called GRPR. This is a 2-part study. Participation could last up to 36 weeks or until your tumor progresses.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically proven diagnosis of locally advanced, unresectable, or metastatic cancer.
* Must be assessed by computed tomography (CT)/magnetic resonance imaging (MRI) to confirm at least 1 of the following:

  * At least 1 measurable target lesion per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
  * If only bone lesions are present without a soft-tissue component, a bone scan or MRI must confirm at least 2 detectable lesions considered to represent active metastases
* Must have GRPR-positive disease, defined by investigator assessment of GRPR imaging.
* Must have the following histologically or cytologically confirmed diagnosis:

  * Estrogen receptor (ER+)/human epidermal growth factor receptor 2 (HER2-) breast cancer
  * ER+/HER2+ breast cancer
  * Colorectal carcinoma
  * Metastatic castration-resistant prostate cancer
  * Endometrial carcinoma. Carcinosarcoma is eligible. Uterine leiomyosarcoma, adenosarcoma, or endometrial stromal sarcoma is not eligible.
  * Other GRPR-positive solid tumor
* For participants with breast cancer diagnosis, where possible, ER and HER2 status should be assessed from the most recent tissue biopsy taken at the time of presentation with recurrent or metastatic disease.

  * To fulfill the requirement for ER+ disease by local testing, a tumor must express the ER immunohistochemistry, as defined in the relevant American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
  * HER2 status should be determined by local testing, as defined in the relevant ASCO/CAP Guidelines.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 1.
* Must be able to comply with outpatient treatment, laboratory monitoring, imaging, and required clinic visits for the duration of trial participation.

Exclusion Criteria:

* Phase 1a (Cohort A1 and A2) only: Previously received radiopharmaceutical or radioligand therapy. For participants with metastatic castration-resistant prostate cancer (mCRPC), prior ¹⁷⁷Lu-prostate-specific membrane antigen (PSMA)-617 is permitted.
* Has a history of ongoing acute pancreatitis within 1 year of screening.
* Previously received any prior hemi-body or whole-body radiotherapy, or prior external beam radiation therapy (EBRT) to greater than 25% of the bone marrow.
* A bone superscan, defined as a bone scan that demonstrates markedly increased skeletal radioisotope uptake relative to soft tissues in association with absent or faint genitourinary tract activity.
* Has evidence of ongoing and untreated urinary tract obstruction or unmanageable urinary incontinence.
* Have known active hepatitis B virus (HBV) defined as positive for hepatitis B surface antigen (HBsAg) or Polymerase Chain Reaction (PCR) positive for HBV deoxyribonucleic acid (DNA) . Exception: Individuals with chronic HBV if they:

  * Have positive HBsAg
  * Are on suppressive antiviral therapy, as allowed per local regulations prior to C1D1
  * Remain on the same antiviral treatment throughout study, and should follow local standards for continuation of therapy after completion of trial therapy.
  * Have undetectable HBV DNA ≤14 days of C1D1.
* Have known active hepatitis C virus (HCV) defined as positive for anti-HCV antibodies. Exception: Individuals previously treated for HCV if they:

  * Completed curative antiviral therapy.
  * Have an HCV viral load below the limit of quantification ≤14 days of C1D1 and.
  * Are positive for anti-HCV antibodies and negative for HCV ribonucleic acid (RNA) before randomization.
* Have untreated human immunodeficiency virus (HIV) infection. Exception: Individuals who have well-controlled HIV infection/disease and they:

  * Are on a stable and permitted antiretroviral therapy (ART) regimen without changes in drug or dose, for at least 4 weeks prior to C1D1
  * Have a viral load of <400 copies/mL ≤14 days of C1D1.
  * Have a CD4+ T-cell count ≥350 cells/mL ≤14 days of C1D1.
  * Have not had an opportunistic infection within the past 12 months.
* Has an active second malignancy unless in remission with life expectancy greater than 2 years.
* Has known hypersensitivity to any component or excipient of LY4257496.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Phase 1a Dose Escalation: Maximum Tolerated Dose of LY4257496 | From Cycle 1 Day 1 (C1D1) through 28 days after the first dose of study drug. Cycle = 28 days
Phase 1a Dose Optimization: Number of Dose Limiting Toxicities of LY4257496 | From Cycle 1 Day 1 (C1D1) through 28 days after the first dose of study drug. Cycle = 28 days
Phase 1b Dose Expansion and Optimization: Objective Response Rate (ORR): Percentage of Participants with Best Response of Complete Response (CR) or Partial Response (PR) | From C1D1 through efficacy follow-up, estimated as Week 42. Cycle = 42 weeks

SECONDARY OUTCOMES:
Phase 1a Dose Escalation and Optimization: ORR: Percentage of Participants with Best Response of CR or PR | From C1D1 through efficacy follow-up, estimated as Week 42. Cycle = 42 weeks
Phase 1a Dose Escalation: Absorbed Dose Estimates (Gray (Gy)) of LY4257496 in Normal Organs | From C1D1 through 30 days after the last dose of study drug dose. Cycle = 30 days
Phase 1a Dose Escalation and Optimization: Absorbed Dose Estimates (Gy) of LY4257529 in Normal Organs | From end of injection at Screening, and at Day 30 through 1 day after injection
Phase 1a Dose Escalation Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of LY4257496 | From C1D1 through 30 days after the last dose of study drug dose. Cycle = 30 days
Phase 1a Dose Escalation and Optimization PK: Cmax of LY4257529 | From end of injection through 1 day after injection
Phase 1a Dose Escalation PK: Area Under the Curve (AUC) of LY4257496 | From C1D1 through 30 days after the last dose of study drug dose. Cycle = 30 days
Phase 1a Dose Escalation and Optimization PK: AUC of LY4257529 | From end of injection through 1 day after injection

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- United States (14):
  - City of Hope, Duarte, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Biogenix Molecular, LLC, Miami, Florida
  - Moffitt, Tampa, Florida
  - Emory University School of Medicine - Winship Cancer Institute, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - BAMF Health Inc., Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Texas Oncology - DFW (Sammons CC), Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Canada (4):
  - Juravinski Cancer Centre, Hamilton
  - Lady Davis Institute for Medical Research Jewish General Hospital, Montreal
  - Sunnybrook Health Sciences Centre, Toronto
  - Princess Margaret Hospital, Toronto
- France (2):
  - Institut Curie, Paris
  - Institut de Cancerologie de l'Ouest - site St-Herblain, Saint-Herblain
- Germany (3):
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - LMU Klinikum Muenchen-Campus Grosshadern, München
- Hospital Universitari Quiron Dexeus Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY4257496 in Participants With Cancer (OMNIRAY) — https://trials.lilly.com/en-US/trial/637755